CLINICAL TRIAL: NCT07019805
Title: Risk Factors for Post-Induction Hypotension Following General Anesthesia in Geriatric Patients Undergoing Elective Non-Cardiac Surgery : A Prospective Study
Brief Title: What Causes Low Blood Pressure After Anesthesia in Older Adults Having Non-Heart Surgery ?
Acronym: GERIHYPO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Dr. dr. Aida Rosita Tantri, Sp.An-TI, Subsp. AR (K), Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-08-1341
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Geriatric; General Anesthesia Induced Hypotension; Elective Surgery; Hypotension; Risk Factor
Keywords: Geriatric; Hypotension; General Anesthesia; Risk Factor
MeSH Terms: conditions — Hypotension | interventions — Fentanyl; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Geriatric Patients Receiving General Anesthesia for Elective Non-Cardiac Surgery (Other): This arm includes geriatric patients (aged 60 years and older) undergoing elective non-cardiac surgery under general anesthesia. The study will observe and record the occurrence of post-induction hypotension and evaluate various patient-related and anesthesia-related risk factors that may contribute to its development. No experimental intervention will be administered as this is an observational study.
  Interventions: Drug: Standard General Anesthesia Induction Using Propofol, Fentanyl and Midazolam; Device: Blood Pressure Continous Monitoring, syrnge pump for the anesthesia agent, and vasoconstrictor drug

INTERVENTIONS:
Drug: Standard General Anesthesia Induction Using Propofol, Fentanyl and Midazolam — This intervention refers to the standard induction of general anesthesia in geriatric patients undergoing elective non-cardiac surgery. Induction typically involves the administration of intravenous anesthetic agents such as propofol and fentanyl, based on institutional protocols and the anesthesiologist's discretion. This study does not modify or introduce any new treatment; it merely observes and records peri-induction parameters to identify factors associated with the occurrence of post-induction hypotension.
Device: Blood Pressure Continous Monitoring, syrnge pump for the anesthesia agent, and vasoconstrictor drug — This intervention involves the standard clinical use of non-invasive continuous blood pressure monitoring during the induction of general anesthesia in geriatric patients undergoing elective non-cardiac surgery. Intravenous anesthetic agents (e.g., propofol, fentanyl) and vasopressors (e.g., ephedrine, norepinephrine) are administered via syringe pumps based on the anesthesiologist's clinical judgment. The study does not introduce any experimental treatment but observes blood pressure changes in real time to identify risk factors for post-induction hypotension. The integration of continuous hemodynamic monitoring distinguishes this observational approach from routine anesthetic induction without such monitoring.

SUMMARY:
The purpose of this study is to identify risk factors contributing to post-induction hypotension in geriatric patients undergoing elective non-cardiac surgery under general anesthesia at Dr. Cipto Mangunkusumo National Central Public Hospital. Post-induction hypotension is defined as a decrease in Mean Arterial Pressure (MAP) of more than 30% from baseline after anesthesia induction up to 20 minutes post-induction. This condition can lead to adverse effects such as myocardial injury, acute kidney injury, stroke, and even death.

This research aims to answer several key questions, including whether the following factors influence the risk of post-induction hypotension:

* Airway management with endotracheal intubation.
* Low albumin levels.
* Presence of comorbidities such as hypertension, cancer/malignancy, diabetes mellitus, chronic heart disease, and chronic kidney failure.
* Dose of propofol during anesthesia induction.
* Dose of fentanyl administered during anesthesia induction.
* Dose of midazolam administered during anesthesia induction.
* Frailty score.

This study is an observational analytical study with a prospective cohort design. Data will be collected from medical records and direct observation of geriatric patients who meet the inclusion and exclusion criteria. Sampling will be done using a consecutive sampling method. The targeted sample size is 333 subjects, accounting for a 10% dropout rate.

Study subjects will meet the inclusion criteria: geriatric patients over 60 years old undergoing elective non-cardiac surgery under general anesthesia with ASA (American Society of Anesthesiologists) classification I-IV. Exclusion criteria include patients receiving a combination of general anesthesia with regional or epidural anesthesia, more than 2 attempts at endotracheal intubation, patients already intubated before the surgical procedure, those receiving vasopressors or inotropics before general anesthesia induction, and intentional hypotension within 20 minutes after intubation.

The data to be recorded include patient characteristics, ASA classification, history of comorbidities, medications consumed, vital signs (before entering the operating room, upon arrival in the operating room, immediately after intubation, and at 5, 10, 15, and 20 minutes after intubation), type of surgery, anesthesia technique, type of anesthetic gas used, total doses of propofol, fentanyl, and midazolam with their administration times, laboratory results, chest X-ray results, presence or absence of endotracheal intubation procedure, administration of vasopressors or inotropics before induction, and patient position during blood pressure measurements. Data analysis will be performed using Graphpad Prism version 10 for MacOS, including descriptive analysis, normality tests, bivariate tests (Chi-square or Fisher's exact test, T-test or Mann-Whitney), and multivariate analysis using Cox regression to identify risk factors and determine relative risk.

DETAILED DESCRIPTION:
Research Title: Risk Factors for Post-Induction Hypotension in Geriatric Patients Undergoing Elective Non-Cardiac Surgery Under General Anesthesia

Researcher: Dr. dr. Aida Rosita Tantri, Sp.An-TI, Subsp.An.R (K)

Institution: Department of Anesthesiology and Intensive Therapy, Faculty of Medicine, University of Indonesia, Jakarta, 2024

Background:

General anesthesia aims to achieve the anesthetic triad: loss of consciousness, loss of pain, and skeletal muscle relaxation. However, general anesthesia can also cause adverse effects, one of which is hemodynamic instability like hypotension. Hypotension is the most commonly encountered hemodynamic disturbance and can occur immediately after the completion of general anesthesia induction until the start of surgery. Post-induction hypotension carries a risk of adverse conditions such as myocardial injury, acute kidney injury, stroke, and mortality. The definition of hypotension varies, with incidence ranging from 5-99%. Some definitions mentioned include systolic blood pressure <90 mmHg or receiving at least one norepinephrine infusion at a rate of >6 micrograms (mcg) per minute within 20 minutes post-induction (Südfeld et al.), as well as a decrease in Mean Arterial Pressure (MAP) of more than 30% compared to baseline or initial data (Jor et al. and Bijker et al.). Perioperative morbidity is more frequent in the geriatric age group, making increasing age one of the predictive factors for post-induction hypotension. Other risk factors that have been studied include hypertension upon arrival in the operating room, increased fentanyl dosage, induction with propofol, and the degree of frailty. By understanding these risk factors, it is hoped that complications from post-induction hypotension can be prevented.

Problem Statement:

Post-induction hypotension in general anesthesia, characterized by a decrease in MAP >30% compared to baseline MAP, is a common complication with extensively described negative effects. Although various factors have been studied to predict the occurrence of post-anesthesia hypotension, specific studies on geriatric patients undergoing elective non-cardiac surgery under general anesthesia have not yet been conducted in Indonesia, particularly at Dr. Cipto Mangunkusumo National Central Public Hospital.

Research Questions:

* Does airway management with endotracheal intubation affect the risk of post-induction hypotension in geriatric patients undergoing non-cardiac surgery?
* Does a low albumin level affect the risk of post-induction hypotension in geriatric patients undergoing non-cardiac surgery?
* Does the presence of comorbid diseases (hypertension, cancer/malignancy, diabetes mellitus, chronic heart disease, chronic kidney failure) affect the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery?
* Does the dose of propofol during anesthesia induction affect the risk of post-induction hypotension in geriatric patients undergoing non-cardiac surgery?
* Does the dose of fentanyl administered during anesthesia induction affect the risk of post-induction hypotension in geriatric patients undergoing non-cardiac surgery?
* Does the dose of midazolam administered during anesthesia induction affect the risk of post-induction hypotension in geriatric patients undergoing non-cardiac surgery?
* Does the frailty score affect the risk of post-induction hypotension in geriatric patients undergoing non-cardiac surgery?

Research Hypotheses:

* Airway management with endotracheal intubation affects the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery.
* Low albumin levels affect the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery.
* The presence of comorbid diseases (hypertension, dyslipidemia, cancer, diabetes mellitus, chronic heart disease, chronic kidney failure) affects the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery.
* The dose of propofol during induction affects the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery.
* The dose of fentanyl during induction affects the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery.
* The dose of midazolam during induction affects the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery.
* The frailty score affects the risk of post-induction hypotension in geriatric patients undergoing non-cardiac surgery.

Research Objectives:

* General Objective: To identify risk factors for post-induction hypotension in geriatric patients undergoing non-cardiac surgery under general anesthesia at Dr. Cipto Mangunkusumo National Central Public Hospital.
* Specific Objectives:

  * To analyze the relationship between airway management and the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery under general anesthesia.
  * To analyze the relationship between albumin levels and the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery under general anesthesia.
  * To analyze the relationship between comorbid diseases and the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery under general anesthesia.
  * To analyze the relationship between propofol dose during induction and the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery under general anesthesia.
  * To analyze the relationship between fentanyl dose and the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery under general anesthesia.
  * To analyze the relationship between midazolam dose and the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery under general anesthesia.
  * To analyze the relationship between frailty score and the incidence of post-induction hypotension in geriatric patients undergoing non-cardiac surgery under general anesthesia.

Research Benefits:

The results of this study are expected to provide useful information for researchers, educational institutions, and public services. By identifying risk factors for post-induction hypotension, it is hoped that this can serve as a basis for prevention efforts, minimization, and appropriate management of the negative effects of post-induction hypotension, especially for the geriatric population undergoing general anesthesia. For educational institutions, this research will add information and knowledge to predict and minimize the negative effects of post-induction hypotension. For the community, it is expected to provide information and education about risk factors for post-induction hypotension, especially for geriatrics undergoing surgery with general anesthesia. For researchers, these results can serve as a basis and reference for further research development, as well as contribute knowledge on risk factors for post-induction hypotension in geriatric patients undergoing non-cardiac surgery.

Research Methodology:

* Research Design: Observational analytic study with a prospective cohort design.
* Location and Time of Research: Kanigara and Kirana operating theaters at Dr. Cipto Mangunkusumo National Central Public Hospital, estimated to be from September 2024 to March 2025.
* Population and Sample:

Target Population: All geriatric patients undergoing elective non-cardiac surgical procedures under general anesthesia at Dr. Cipto Mangunkusumo National Central Public Hospital.

* Inclusion Criteria: Geriatric patients aged over 60 years undergoing elective non-cardiac surgical procedures under general anesthesia, with ASA (American Society of Anesthesiologists) classification I-IV.
* Exclusion Criteria: Patients receiving a combination of general anesthesia with regional or epidural anesthesia, more than 2 attempts at endotracheal intubation, patients already intubated before the surgical procedure, those receiving vasopressors or inotropic infusions before general anesthesia induction, and intentional hypotension within 20 minutes after intubation.
* Sample Size Estimation: Calculated using sample formulas for comparing two proportions (Jor et al., Kawasaki et al., Green et al., Lee et al. ) and a rule of thumb formula. Based on calculations using the individual factor risk formulas, the largest sample size required for each variable is 100 subjects, resulting in a total of 200 subjects for both groups. Considering a 10% dropout rate, the total sample required is 220 subjects. However, using the "rules of thumb" formula, a total sample of 303 subjects is obtained for both groups, and with a 10% dropout rate, the total sample becomes 333 subjects. Therefore, the total number of subjects in this study will be 333.

Research Procedure:

* Research Instruments: Patient data collection form (CRF) to record patient characteristics, ASA classification, history of comorbid diseases, medications consumed, vital signs (before entering the operating room, upon arrival in the operating room, immediately after intubation, and at 5, 10, 15, 20 minutes after intubation), type of surgery, anesthesia technique, type of anesthetic gas used, total doses of propofol, fentanyl, and midazolam with their administration times, laboratory results, chest X-ray results, presence or absence of endotracheal intubation procedure, administration of vasopressors or inotropics before induction, and patient position during blood pressure measurements.
* Subject Recruitment: Begins after ethical approval from KEPK FKUI - RSCM and permission from the director of Dr. Cipto Mangunkusumo National Central Public Hospital have been issued. Subjects meeting the inclusion and exclusion criteria will be used as study samples. An explanation of the study's purpose, procedures, benefits, and risks will be provided to the patient or accompanying family members, followed by the signing of an informed consent form. Sample collection will be done through consecutive sampling.
* Research Implementation: Data from medical records will be copied into the research form (CRF) and then transferred into a Microsoft Excel soft file for data tabulation.

Research Variables:

* Dependent Variable: Post-induction hypotension.
* Independent Variables: Airway management, albumin levels, comorbid diseases (hypertension, diabetes mellitus, cancer/malignancy, chronic cardiac disease, chronic kidney failure), propofol use and dose, fentanyl use and dose, and midazolam use and dose.

Operational Definition: Detailed definitions and methods of measurement for each variable (gender, age, BMI, ASA classification, post-induction hypotension, airway management, albumin levels, comorbid diseases, pulse rate, MAP before and after induction, T0, TEI, T5, T10, T15, T20, propofol dose, fentanyl dose, midazolam dose, frailty score) are presented in a table.

Data Analysis: Analysis will be performed using Graphpad Prism version 10 for MacOS. The analysis stages include descriptive analysis, normality testing (Kolmogorov Smirnov test), presentation of categorical data (counts and percentages), and numerical data (mean ± standard deviation for normally distributed data, and median (min - max) for non-normally distributed data). Bivariate analysis will use the Chi-square test or Fisher's exact test for categorical data, and the unpaired T-test or Mann-Whitney test for numerical data. Multivariate analysis will be conducted on variables with a p-value < 0.25 in bivariate analysis using Cox regression to identify determinant risk factors and determine the relative risk. A 95% confidence interval will be used, with a p-value < 0.05 considered statistically significant. Receiver operating characteristic (ROC) curves will be generated to measure the discriminative power of risk factors.

Research Ethics:

Ethical approval for the research will be obtained from the Health Research Ethics Committee of the Faculty of Medicine, University of Indonesia - Dr. Cipto Mangunkusumo National Central Public Hospital. Once ethical approval and research site permits are issued, the research can commence, adhering to ethical principles: autonomy (informed consent from subjects after receiving information on objectives, procedures, benefits, and risks, ensuring confidentiality), justice (subjects will undergo anesthesia as planned, with no changes in technique, and data will only be collected from medical records), beneficence (researchers will ensure subject benefit and comfort during the study), and non-maleficence (transparent reporting to the ethics committee in case of incidents or undesirable events).

ELIGIBILITY:
Inclusion Criteria:

* Geriatric patients aged over 60 years undergoing elective non-cardiac surgical procedures under general anesthesia, with ASA (American Society of Anesthesiologists) classification I-IV.

Exclusion Criteria:

* Patients receiving a combination of general anesthesia with regional or epidural anesthesia, more than 2 attempts at endotracheal intubation, patients already intubated before the surgical procedure, those receiving vasopressors or inotropic infusions before general anesthesia induction, and intentional hypotension within 20 minutes after intubation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Association Between Pre-Induction Risk Factors and Post-Induction Hypotension | Baseline to 20 minutes post-induction
  Hypotension is defined as a decrease in mean arterial pressure (MAP) of more than 20% from baseline or MAP < 65 mmHg within 10 minutes after induction. The study will record the presence or absence of hypotension in each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Kepk Fkui-Rscm, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
All data collected through this study will be kept confidential. The identity of each respondent will be presented only as initials and can only be accessed by the research team and the health research ethics committee for verification purposes. Presentation of the research results at scientific meetings or in any form of scientific publication will not include your name or any personal identifying information.

REFERENCES:
- [Background] Reich DL, Hossain S, Krol M, Baez B, Patel P, Bernstein A, Bodian CA. Predictors of hypotension after induction of general anesthesia. Anesth Analg. 2005 Sep;101(3):622-628. doi: 10.1213/01.ANE.0000175214.38450.91. PMID 16115962
- [Background] Sutthibenjakul K, Chatmongkolchart S. Risk factors for postinduction hypotension among elderly patients undergoing elective non-cardiac surgery under general anesthesia. Journal of Health Science and Medical Research. 2021;39(5).
- [Background] Lim BG, Lee IO. Anesthetic management of geriatric patients. Korean J Anesthesiol. 2020 Feb;73(1):8-29. doi: 10.4097/kja.19391. Epub 2019 Oct 22. PMID 31636241
- [Background] Jor O, Maca J, Koutna J, Gemrotova M, Vymazal T, Litschmannova M, Sevcik P, Reimer P, Mikulova V, Trlicova M, Cerny V. Hypotension after induction of general anesthesia: occurrence, risk factors, and therapy. A prospective multicentre observational study. J Anesth. 2018 Oct;32(5):673-680. doi: 10.1007/s00540-018-2532-6. Epub 2018 Jul 19. PMID 30027443
- [Background] Bijker JB, Persoon S, Peelen LM, Moons KG, Kalkman CJ, Kappelle LJ, van Klei WA. Intraoperative hypotension and perioperative ischemic stroke after general surgery: a nested case-control study. Anesthesiology. 2012 Mar;116(3):658-64. doi: 10.1097/ALN.0b013e3182472320. PMID 22277949
- [Background] de la Hoz MA, Rangasamy V, Bastos AB, Xu X, Novack V, Saugel B, Subramaniam B. Intraoperative Hypotension and Acute Kidney Injury, Stroke, and Mortality during and outside Cardiopulmonary Bypass: A Retrospective Observational Cohort Study. Anesthesiology. 2022 Jun 1;136(6):927-939. doi: 10.1097/ALN.0000000000004175. PMID 35188970
- [Background] Mangku G, Senaphati TGA. Buku ajar ilmu anastesia dan reanimasi. PT Indeks. 2010.
- [Background] Sudfeld S, Brechnitz S, Wagner JY, Reese PC, Pinnschmidt HO, Reuter DA, Saugel B. Post-induction hypotension and early intraoperative hypotension associated with general anaesthesia. Br J Anaesth. 2017 Jul 1;119(1):57-64. doi: 10.1093/bja/aex127. PMID 28974066